CLINICAL TRIAL: NCT05794425
Title: A Multicenter Collaborative Clinical Study of Umbilical Cord Blood Combined With Umbilical Cord Derived Mesenchymal Stem Cells in the Treatment of Bone Marrow Failure Disorders
Brief Title: Clinical Study of UCB Combined With UC-MSCs in the Treatment of Bone Marrow Failure Disorders
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shandong Qilu Stem Cells Engineering Co., Ltd. (Industry)
Collaborators: Shandong Province Third hospital (Other); Dezhou People's Hospital (Other); Children's Hospital Affiliated to Shandong University (Unknown); The Second Affiliated Hospital of Shandong First Medical University (Other); Tai'an Central Hospital (Unknown); Linyi People's Hospital (Other); Rizhao People's Hospital (Other); Lanling People's Hospital (Unknown); Jining First People's Hospital (Other); Jining Medical University (Other); Zibo Municipal Hospital (Other); Binzhou People's Hospital (Other); The Affiliated Hospital of Binzhou Medical College (Unknown); Shengli Oilfield Hospital (Other); Weihai Municipal Hospital (Other); Weihai Central Hospital (Other); Shandong University of Traditional Chinese Medicine (Other); Gansu Provincial Hospital of Traditional Chinese Medicine (TCM) (Unknown); Wuwei People's Hospital (Unknown); Gansu Wuwei Tumor Hospital (Other); The Second Affiliated Hospital of Harbin Medical University (Other); Yuncheng Institute of Hematology (Unknown); Kaifeng Central Hospital (Other); Zhengzhou Central Hospital (Other); Air Force Hospital of Western War Zone (Unknown); The First People' s Hospital of Yunnan Province (Unknown); Zigong No.1 Peoples Hospital (Other); The First People's Hospital of Jingzhou (Other); Jiangxi Province Children's Hospital (Other); Second Affiliated Hospital of Zhengzhou University (Other); Yantai Ludong Hospital (Shandong Provincial Hospital Group) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UCB&MSCs-BMF-2023
Record Dates: First submitted 2023-03-20; First posted 2023-04-03 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Bone Marrow Failure Disorders
MeSH Terms: conditions — Bone Marrow Failure Disorders | interventions — Cyclosporine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cyclosporine A (Experimental)
  Interventions: Drug: Cyclosporine A
- UCB+UC-MSCs (Experimental)
  Interventions: Biological: Umbilical cord blood & Umbilical cord derived mesenchymal stem cells

INTERVENTIONS:
Drug: Cyclosporine A — 3-5 mg per kilogram per day.
  Arms: Cyclosporine A
Biological: Umbilical cord blood & Umbilical cord derived mesenchymal stem cells — Intravenous infusion of umbilical cord blood and umbilical cord derived mesenchymal stem cells (5-8×10^7) at 1 week interval.
  Arms: UCB+UC-MSCs

SUMMARY:
The multicenter collaborative clinical study conducted a systematic clinical observation in the treatment of bone marrow failure diseases via UCB&UC-MSCs , in order to observe its clinical efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with bone marrow failure disorders, including aplastic anemia, pure red cell aplastic anemia, immune-related pancytopenia, paroxysmal nocturnal hemoglobinuria, myelodysplastic syndrome, acute arrest of hemopoiesis, and cytopenia of unknown significance;
2. Patients with no severe impairment of liver and kidney function (total bilirubin (TBIL): ≤ 1.5×ULN; ALT or AST: ≤ 2.5×ULN; Alkaline phosphatase: ≤ 3×ULN; Serum creatinine: ≤ 1.5×ULN);
3. The prothrombin time (PT) or activated partial thrombin time (APTT) or international normalized ratio (INR): ≤ 1.5×ULN in the absence of anticoagulant therapy;
4. The left ventricular ejection fraction (LVEF): ≥50% by cardiac echocardiography
5. Hepatitis B surface antigen (HBsAg) and Hepatitis B core antibody (HBcAb) were negative. If any of the above items is positive, the HBV DNA titer in peripheral blood must be lower than the detection limit or 1×10^3 copys/ml;
6. Patients with no plans for stem cell transplantation;
7. Patients with ECOG 0-2;
8. Those who voluntarily participate in this clinical study and have signed an informed consent .

Exclusion Criteria:

1. Patients who have suffered malignant tumors other than squamous cell carcinoma of the skin, basal cell carcinoma of the skin, malignant melanoma cured by surgery, and carcinoma in situ of the cervix in the past 5 years;
2. Patient with severe cardiac insufficiency (e.g. grade Ⅲ、Ⅳ by NYHA classification NYHA), and medically uncontrolled hypertension (systolic blood pressure ≥ 160 mmHg or diastolic blood pressure ≥110 mmHg);
3. Patients with severe mental illness;
4. Patients with clinically significant infection should be recruited with delay;
5. AST or ALT: above 3 times the upper limit of normal, creatinine, total bilirubin, or alkaline: phosphatase (ALP): above 1.5 times the upper limit of normal;
6. Patients with test positive for HIV, HCV or syphilis;
7. Patients with severe allergies or allergic to the active ingredients, excipients of the drug, or blood products in this clinical trials;
8. Patients who are pregnant or breastfeeding, or have a childbirth plan in the near future;
9. Patients receive allogeneic/autologous hematopoietic stem cell transplantation by the assessment of investigators;
10. There are other conditions that the investigators consider inappropriate for inclusion.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Up to two years
  To evaluate efficacy of UCB in combination with UC-MSCs in the treatment of bone marrow failure disorders

SECONDARY OUTCOMES:
Progression-free Survival (PFS) | Up to two years
  To assess Progression-free Survival (PFS) of the combination
Overall Survival (OS) | Up to two years
  To assess overall survival (OS) of the combination

CONTACTS AND LOCATIONS:
Overall Officials: zhe Yu, MD, Principal Investigator — Shandong Province Third hospital
Locations (8):
- China (8):
  - Shandong Provincial Third Hospital, Jinan, Shandong
  - Affiliated Hospital of Shandong University of Traditional Chinese Medicine, Jinan, Shandong
  - Jining first people's Hospital, Jining, Shandong
  - Linyi People's Hospital, Linyi, Shandong
  - Rizhao People's Hospital, Rizhao, Shandong
  - Tai'an Central Hospital, Tai’an, Shandong
  - Weihai Municipal Hospital, Weihai, Shandong
  - Yantai Ludong Hospital (Shandong Provincial Hospital Group), Yantai, Shandong

IPD SHARING:
Plan to Share IPD: No